CLINICAL TRIAL: NCT01483118
Title: The Effects of Oral Cinnamon Extract on Menstrual Cyclicity in PolyCystic Ovary Syndrome
Brief Title: Cinnamon Extract on Menstrual Cycles in PolyCystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rogerio A. Lobo (Other)
Collaborators: Integrity Nutraceuticals International (Unknown)
Responsible Party: Sponsor-Investigator, Rogerio A. Lobo, Professor of Obstetrics and Gynecology, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAI1377
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; Insulin resistance; Cinnamon extract; Irregular menstrual cycles; Ovarian cysts
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Menstruation Disturbances; Ovarian Cysts | interventions — cinnulin PF

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cinnamon Extract Arm (Active Comparator): PCOS patients receiving abstract of cinnamon
  Interventions: Drug: Cinnamon Extract
- Placebo Arm (Placebo Comparator): PCOS patients receiving placebo capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Cinnamon Extract — Purified aqueous abstract of cinnamon in 125mg capsules, which would be taken orally before each meal, for a total of 1,500mg/day for 6 months.
  Other Names: Cinnulin PF
  Arms: Cinnamon Extract Arm
Dietary Supplement: Placebo — Placebo capsules containing ground cereal.
  Arms: Placebo Arm

SUMMARY:
The primary purpose of this follow-up study is to determine if cinnamon can restore menstrual cyclicity in Polycystic Ovary Syndrome (PCOS) subjects with oligomenorrhea. As a secondary purpose, the investigators intend to confirm the salutatory effect of cinnamon on insulin resistance in larger group of study subjects.

Polycystic ovary syndrome (PCOS) is a very common condition found in women of childbearing age. PCOS patients often have irregular periods, extra hair growth, or difficulty becoming pregnant. The syndrome can also be associated with more serious conditions such as heart disease, diabetes, or cancer of the uterus. Although no one knows the cause of the syndrome, scientific studies showed that having too much insulin can be one of the reasons. In fact, almost every overweight woman with PCOS has been found to have high insulin levels.

Recently studies using rats and mice have shown that a commonly used spice, cinnamon, may also reduce the body's insulin level. Another study showed that daily use of cinnamon for forty days lowered the blood sugar level in patients with diabetes. Our own study also showed that using cinnamon everyday for 8 weeks decreased insulin resistance in women with PCOS. The purpose of this study is to see if cinnamon can help women with PCOS have more regular periods.

DETAILED DESCRIPTION:
All patients will eat a balanced diet containing 1800 calories per day, but half of the patients in the study will take pre-made cinnamon extract pills three times a day, while the other half will take placebo pills (pills with no cinnamon extract) three times a day for 6 months. During this time, every patient will keep track of her period on a calendar.

Blood tests measuring insulin, substances important for insulin action, cholesterol, and glucose (sugar) will be taken before and after the 6 months of medication. A total of 8 separate visits will be needed to finish the study. At the end of the study, the investigators will then compare the number of periods, blood glucose, insulin, and cholesterol levels between the patients that took cinnamon and the patients that took placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged greater than 18 years of age
* Ability to understand and willingness to comply with the study protocol
* Written informed consent
* Patients meeting the Rotterdam PCOS workshop criteria for polycystic ovary syndrome, defined by oligomenorrhea or amenorrhea and at least one of the following two signs: clinical or biochemical evidence of hyperandrogenism or ultrasound finding of polycystic appearing ovaries.

Exclusion Criteria:

* Current pregnancy or lactation
* Liver disease or elevated liver enzymes
* Established diagnosis of diabetes mellitus
* Abnormal serum glucose levels either at fasting or after the 2-hr oral glucose tolerance test meeting criteria for the diagnosis of diabetes mellitus according to the American Diabetes Association.
* Insulin sensitizing treatment within 3 months prior to or during the eight week study period.
* Hormonal treatment involving estrogen or progesterone 3 months prior to or during the study period, with the exception of medroxyprogesterone acetate for withdrawal bleeding.
* Systemic or inhaled corticosteroids.
* Known hypersensitive reaction to cinnamon.
* Patients with seizure disorders, known cardiovascular disease, or cerebrovascular disease.
* Body mass index (BMI)range 20-50 (excluding all women with BMI under 20 or over 50).

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-03; Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Lobo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kort DH, Lobo RA. Preliminary evidence that cinnamon improves menstrual cyclicity in women with polycystic ovary syndrome: a randomized controlled trial. Am J Obstet Gynecol. 2014 Nov;211(5):487.e1-6. doi: 10.1016/j.ajog.2014.05.009. Epub 2014 May 9. PMID 24813595

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Advertizing in newspaper beginning in August 2011
Groups:
- Cinnamon Extract Arm: Purified aqueous abstract of cinnamon in 125mg capsules
  Cinnamon Extract: Purified aqueous abstract of cinnamon in 125mg capsules, which would be taken orally before each meal, for a total of 1,500mg/day for 6 months.
- Placebo Arm: Placebo capsules containing ground cereal.
  Placebo: Placebo capsules containing ground cereal.
Period: Overall Study
Arm/Group | Cinnamon Extract Arm | Placebo Arm
Started | 23 | 22
Completed 3 Months | 15 | 11
Completed ((entire 6 months)) | 11 | 6
Not Completed | 12 | 16
Not completed — Lost to Follow-up | 12 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cinnamon Extract Arm | Placebo Arm | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Continuous [Mean (Full Range); unit: years] | 26.95 [18 to 34] | 27.86 [18 to 38] | 27.5 [18 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 14 | 13 | 27
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Menses During the Six Month Study Period.
Description: Ovulatory cycles will be confirmed by serum progesterone levels.
Time Frame: Up to 6 months
Measure: Median (Inter-Quartile Range); unit: Number of menstrual cycles per month
Groups:
- Cinnamon Extract Arm: Purified aqueous abstract of cinnamon in 125mg capsules
  Cinnamon Extract: Purified aqueous abstract of cinnamon in 125mg capsules, which would be taken orally before each meal, for a total of 1,500mg/day for 6 months.
  Baseline (no. of cycles/month) 0.42 Study period (no. of cycles/month) 0.75 Change during study +/- cycles/month +0.23
- Placebo Arm: Placebo capsules containing ground cereal.
  Placebo: Placebo capsules containing ground cereal.
  Baseline (no. of cycles/month) 0.42 Study period (no. of cycles/month) 0.25 Change during study +/- cycles/month -0.13
Arm/Group | Cinnamon Extract Arm | Placebo Arm
Number analyzed (Participants) | 11 | 6
Number of menstrual cycles per month
  Baseline | .42 [.33 to .63] | .42 [.29 to .68]
  Study Period | .75 [.5 to .83] | .25 [0 to .54]

2. Secondary Outcome: Change in Insulin Resistance
Description: The changes in insulin resistance parameters in overweight patients with PCOS between baseline and after 6 months of daily cinnamon compared to the corresponding change in patients receiving 6 months of placebo. Higher values of insulin resistance represent a worse outcome. A higher value Homeostasis Model of Insulin Resistance indicates more insulin resistance so higher values are worse outcomes (a score of >2 is considered healthy for adults with scores >5 being considered severe insulin resistance). For the Quant. Insulin Sensitivity Check Index, a lower value indicates more insulin resistance so lower values are worse outcomes (values can range from .45, which is considered normal in health individuals and .30, which is characteristic of diabetes).
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: Insulin sensitivity indices
Arm/Group | Cinnamon Extract Arm | Placebo Arm
Number analyzed (Participants) | 11 | 6
Insulin sensitivity indices
  Homeostasis Model of Insulin Resistance - Baseline | 2.3 [1.4 to 2.8] | 1.8 [.71 to 3.3]
  Homeostasis Model of Insulin Resistance - 6 months | 2.5 [.97 to 3.3] | 1.2 [.78 to 2.6]
  Quant. Insulin Sensitivity Check Index - Baseline | .34 [.33 to .36] | .35 [.32 to .41]
  Quant. Insulin Sensitivity Check Index - 6 months | .33 [.32 to .39] | .37 [.33 to .40]

3. Secondary Outcome: Change in Glucose Response
Description: Change in Glucose Response - area under the curve (AUC), trapezoidal method - in overweight patients with PCOS between baseline and after 6 months of daily cinnamon compared to the corresponding change in patient receiving 6 months of placebo. Fasting blood samples were drawn followed by a 2 hour glucose tolerance test with blood draws at 30, 60, and 120min post glucose ingestion.
Time Frame: Baseline and 6 Months - fasting bloods, followed by glucose tolerance test with draws at 30, 60, and 120 minutes post glucose ingestion
Measure: Median (Inter-Quartile Range); unit: mg/dL*min
Arm/Group | Cinnamon Extract Arm | Placebo Arm
Number analyzed (Participants) | 11 | 6
mg/dL*min
  Glucose Response (Area under curve) - Baseline | 16,485 [13,995 to 18,964] | 13,298 [11,993 to 15,285]
  Glucose Response (Area under curve) - 6 months | 16,515 [15,068 to 20,190] | 15,420 [14,468 to 17,798]

ADVERSE EVENTS:
Groups:
- Cinnamon Extract Arm: PCOS patients receiving extract of cinnamon
  Cinnamon Extract: Purified aqueous abstract of cinnamon in 125mg capsules, which would be taken orally before each meal, for a total of 1,500mg/day for 6 months.
Arm/Group | Cinnamon Extract Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/22
Other Adverse Events (participants affected / at risk) | 15/23 | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cinnamon Extract Arm (N=23) | Placebo Arm (N=22)
Right leg swelling with pain (General disorders) | 1 (1) | 0 (0) — Hospitalized
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cinnamon Extract Arm (N=23) | Placebo Arm (N=22)
Acid reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anxiety (General disorders) | 1 (1) | 0 (0)
Back pain (General disorders) | 3 (11) | 1 (1)
Bodyache (General disorders) | 1 (1) | 0 (0)
Breast tenderness (General disorders) | 0 (0) | 1 (1)
Bruise on thigh (General disorders) | 1 (1) | 0 (0)
Bunion (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cold (General disorders) | 3 (6) | 1 (1)
Congestion (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (4) | 0 (0)
Menstrual cramps (Reproductive system and breast disorders) | 6 (7) | 3 (7)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enlarged breast (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Feet swelling (General disorders) | 1 (1) | 0 (0)
Hands/palms swelling (General disorders) | 1 (1) | 0 (0)
Hangover (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 10 (34) | 9 (10)
Heartburn (Gastrointestinal disorders) | 3 (19) | 0 (0)
Heightened sense of smell (General disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Lightheadedness (General disorders) | 1 (1) | 0 (0)
Migraine (General disorders) | 2 (4) | 1 (1)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Nasal congestion (General disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 3 (9) | 1 (1)
Overdose (General disorders) | 0 (0) | 1 (1) — 1 extra dose taken
Pain (General disorders) | 1 (1) | 0 (0) — Due to stomachache
Pink eye (Eye disorders) | 0 (0) | 1 (1) — Right eye affected
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Itchy rash (General disorders) | 1 (1) | 0 (0) — Due to bed bugs
Sleep problem (General disorders) | 0 (0) | 1 (1)
Sleepiness (General disorders) | 0 (0) | 1 (1)
Sore throat (General disorders) | 1 (1) | 1 (1)
Stomachache (General disorders) | 3 (5) | 0 (0)
Stomach cramps (General disorders) | 1 (1) | 0 (0)
Swelling of face (cheeks) (General disorders) | 1 (1) | 0 (0)
Stye in eye (Eye disorders) | 0 (0) | 1 (1)
Swelling of feet and hands (General disorders) | 1 (1) | 0 (0)
Swelling of lips (General disorders) | 1 (1) | 0 (0)
Swelling/puffiness of eye area (General disorders) | 1 (1) | 0 (0)
Throat/nasal congestion (General disorders) | 1 (1) | 0 (0)
Tiredness (General disorders) | 1 (7) | 1 (1)
Toothache (General disorders) | 1 (1) | 1 (1)
Trouble falling asleep (General disorders) | 0 (0) | 1 (2)
Upset stomach (Gastrointestinal disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
High percentage of patients lost to follow up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No